CLINICAL TRIAL: NCT06699043
Title: Comparative Study of Two Different Putty Bone Grafts in Treatment of Intrabony Defects with the Aid of Intramarrow Penetration Technique (Clinical, Radiographical and Histological Evaluation)
Brief Title: Study of Two Different Putty Bone Grafts in Treatment of Intrabony Defects with the Aid of Intramarrow Penetration Technique
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afaf Mansour Dao Abdelslam (Other)
Responsible Party: Sponsor-Investigator, Afaf Mansour Dao Abdelslam, principle investigator, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M0104023OM
Record Dates: First submitted 2024-11-12; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Intrabony Defects in Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: A total of twenty patients will be diagnosed with stage III grade B periodontitis according to the Caton classification. They will be selected from the clinic of Department of Periodontology and Oral Medicine, Faculty of Dentistry, Mansoura University
  Patients will be classified into two groups:
  * Group I: in this group, ten patients with intrabony defect will be treated by open flap debridement with decortication followed by placement of nanocrystalline hydroxyapatite in putty form as grafting material.
  * Group II: in this group, ten patients with intrabony defect will be treated by open flap debridement with decortication followed by placement of Demineralized Bone Matrix allograft putty as grafting material.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nanocrystalline hydroxyapatite in putty form (Active Comparator): • Group I: in this group, ten patients with intrabony defect will be treated by open flap debridement with decortication followed by placement of nanocrystalline hydroxyapatite in putty form as grafting material.
  Interventions: Procedure: nanocrystalline hydroxyapatite in putty form
- Demineralized Bone Matrix allograft putty as grafting material (Active Comparator): group II in this group, ten patients with intrabony defect will be treated by open flap debridement with decortication followed by placement of Demineralized Bone Matrix allograft putty as grafting material.
  Interventions: Procedure: Demineralized Bone Matrix allograft putty

INTERVENTIONS:
Procedure: nanocrystalline hydroxyapatite in putty form — decortication will be performed by penetrating the cortical walls of the intrabony defect by using a round carbide bur of 0.2 mm diameter to reach the marrow space.
  * Multiple perforations will performed not closer than 1mm from each other and deep enough to obtain bleeding from the spongiosa
  * The intrabony defects in Group I will be received nanocrystalline hydroxyapatite in putty form as grafting material (NanoBone® SBX Putty).
  Other Names: guidede tissue regeneration
  Arms: nanocrystalline hydroxyapatite in putty form
Procedure: Demineralized Bone Matrix allograft putty — decortication will be performed by penetrating the cortical walls of the intrabony defect by using a round carbide bur of 0.2 mm diameter to reach the marrow space. • Multiple perforations will performed not closer than 1mm from each other and deep enough to obtain bleeding from the spongiosa • The intrabony defects in Group II will be received Demineralized Bone Matrix allograft putty as grafting material, in both groups will be use membrane to cover of the graft materials and finally will be sutured the flap.
  Arms: Demineralized Bone Matrix allograft putty as grafting material

SUMMARY:
to evaluate and compare efficacy of two different putty forms for both Demineralized Bone Matrix allograft (DBM) and nanocrystalline hydroxyapatite (NCHA) in treatment of intrabony defects with the aid of intramarrow penetration,

A total of twenty patients will be diagnosed with stage III grade B periodontitis according to the Caton classification. They will be selected from the clinic of Department of Periodontology and Oral Medicine, Faculty of Dentistry, Mansoura University

Patients will be classified into two groups:

* Group I: in this group, ten patients with intrabony defect will be treated by open flap debridement with decortication followed by placement of nanocrystalline hydroxyapatite in putty form as grafting material.
* Group II: in this group, ten patients with intrabony defect will be treated by open flap debridement with decortication followed by placement of Demineralized Bone Matrix allograft putty as grafting material.

Clinical assessment:

including the following parameters:

1. Plaque Index (PI).
2. Gingival Index (GI).
3. Clinical Attachment Level (CAL)
4. Probing Depth (PD) Radiological parameters

   * The height of the defect: Distance from the CEJ to the alveolar crest (AC)
   * Depth of the defect: Distance from CEJ to the base of the defect
   * Width of the defect: Highest point of the AC to the root adjacent to the defect
   * Defect angle: Two lines that represent the root surface of the involved tooth and the bone defect surface

DETAILED DESCRIPTION:
Inclusion criteria:

Both genders with 25-55 years of age. Patients with intrabony defects in the Stage III Grade B periodontitis. Individuals with probing depth ≥ 5mm. Individuals with clinical attachment loss ≥ 5mm. Presence of at least one or more intrabony defect ≥ 3 mm on the radiograpgh patients who had not periodontal therapy in the previous 6 months.

Exclusion criteria:

Patient with stage I, II and IV periodontitis. Pregnant or lactating mothers. Patients having any systemic disease. allergies to Local anesthesia and chlorhexidine, antibiotics, and analgesics will be excluded.

Clinical assessment:

including the following parameters: Plaque Index according to Silness P. Loe H 1964. 2. Gingival Index according Loe Silness 1963. 3. Probing pocket depth (PPD) is measured from the free gingival margin to the base of the pocket. 4. Clinical attachment level (CAL) is measured from the cement enamel junction to the base of the pocket.

• In patients All clinical assessments will be recorded at the baseline (immediate before surgery) and after 3 ,6 and 12months post-surgery and radiographic assessments will be recorded at the baseline and after 6 and 12months post-surgery.

This study was conducted following guidelines regulating research work on human subjects of the Faculty of Dentistry, Mansoura University, and the study protocol was reviewed and approved by the Research Ethics Committee of the Faculty of Dentistry, Mansoura University, Egypt. (Number:M0104023OM) All study subjects will sign written informal consent form before enrollment.

Materials:

1. nanocrystalline hydroxyapatite in putty form (NanoBone® SBX Putty) is a unique and patented advanced bone grafting material. It incorporates nano-crystalline particles of hydroxyapatite (HA) that are similar in size, chemistry, and morphology to HA particles occurring in human bone. It is Synthetic biodegradable bone graft substitute consisting of non-sintered nanocrystalline hydroxyapatite in a porous silica gel matrix embedded in an aqueous gel
2. Demineralized Bone Matrix allograft (DBM Putty). presurgical phase:

   * Patients informed consents will be obtained prior to any periodontal treatment.
   * Initial therapy includes full mouth supra and subgingival debridement using ultrasonic scalers and curettes
   * and oral hygiene instruction will be given to all patients in the form of tooth brushing instructions and the use of chlorhexidine mouth wash 2 time daily for 2 weeks.
   * After 4 weeks of initial therapy, all patients will be evaluated to ensure the behavior fitness for periodontal surgery.

surgical phase:

* Prior to surgery all patients will be given pre surgical rinse of 0.2 % Chlorhexidine for 30 seconds.
* The operative site will be anaesthetized using local anesthesia, Buccal and lingual crevicular incisions will be made.
* mucoperiosteal flaps will be reflected, the defect will be thoroughly debridement and root planning will be performed.
* The surgical area will be carefully irrigated with saline and root biomodification will be done.
* For both groups, decortication will be performed by penetrating the cortical walls of the intrabony defect by using a round carbide bur of 0.2 mm diameter to reach the marrow space.
* Multiple perforations will performed not closer than 1mm from each other and deep enough to obtain bleeding from the spongiosa
* The intrabony defects in Group I will be received nanocrystalline hydroxyapatite in putty form as grafting material (NanoBone® SBX Putty).
* Group II will be treated similarly as Group I and the same surgical protocol will followed except that the intrabony defects will be received Demineralized Bone Matrix allograft putty as grafting material, in both groups will be use membrane to cover of the graft materials and finally will be sutured the flap.

post-surgical phase:

* Non-steroidal anti-inflammatory drug and antibiotics will be prescribed.
* chlorhexidine digluconate rinses (0.12%) twice daily for 2 weeks.
* Patients will be advised to consume only soft food during the first week.
* After this period, patients will be reinstructed in mechanical cleaning of the treated teeth using a soft toothbrush and roll technique of brushing for 1 month.
* Sutures will be removed 10 days post operatively. All the patients will be recalled at 3, 6 and 12 months for periodic rechecking.

Statistical Analysis:

All data will be calculated and analyzed by suitable statistical tests

ELIGIBILITY:
Inclusion Criteria:

* Both genders with 25-55 years of age.
* Patients with intrabony defects in the Stage III Grade B periodontitis.
* Individuals with probing depth ≥ 5mm.
* Individuals with clinical attachment loss ≥ 5mm.
* Presence of at least one or more intrabony defect ≥ 3 mm on the radiographs.
* patients who had not periodontal therapy in the previous 6 months.

Exclusion Criteria:

* Patient with stage I, II and IV periodontitis.
* Pregnant or lactating mothers.
* Patients having any systemic disease.
* allergies to Local anesthesia and chlorhexidine, antibiotics, and analgesics will be excluded.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Clinical (Clinical attachment level CAL) | 3,6,12 months
  It was measured since the CEJ to the base of the pocket with UNC-15 periodontal probe
Radiographical Analysis of bone defect | at baseline, 6, 12 months
  Assessment of bone defect area by digital intraoral periapical (IOPA) radiographs.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
it will be decided during the publication times as it may be provided as supplementary files